CLINICAL TRIAL: NCT05713721
Title: SensoMo-PD: Sensorimotor Integration in Monogenic Parkinson-dystonia Syndromes
Brief Title: Sensorimotor Integration in Monogenic Parkinson-dystonia Syndromes
Acronym: SensoMo-PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Anne Weißbach, MD, University Hospital Schleswig-Holstein
Other Study IDs: MJFF-022062
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Parkinson; Dystonia; DYT3; DYT5; PINK1 Gene Deletion; Dystonia, Familial
Keywords: Dystonia; Parkinson's; Parkinson-dystonia; GCH1; Parkin; PINK1; TAF1; XDP; X-linked Dystonia-Parkinsonism
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Parkinson Disease; Dystonia 3, Torsion, X-Linked | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- SMC DYT/PARK-TAF1: Symptomatic mutation carriers (SMC) of the TAF1 gene, which is associated with X-linked Dystonia-Parkinsonism, will be examined.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Other: Video-based clinical examination; Other: 24 hours drug withdrawal of dopaminergic medication; Other: Evaluation of deep brain stimulation
- AMC DYT/PARK-TAF1: Asymptomatic mutation carriers (AMC) of the TAF1 gene will be examined.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Other: Video-based clinical examination
- SMC DYT/PARK-GCH1: Symptomatic mutation carriers (SMC) of the GCH1 gene, which is associated with dopa-responsive Dystonia, will be examined.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Other: Video-based clinical examination; Other: 24 hours drug withdrawal of dopaminergic medication
- AMC DYT/PARK-GCH1: Asymptomatic mutation carriers (AMC) of the GCH1 gene will be examined.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Other: Video-based clinical examination
- SMC PARK-Parkin/PARK-PINK1: Symptomatic mutation carriers (SMC) of the Parkin or PINK1 genes, which is associated with Parkinsonism, will be examined.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Other: Video-based clinical examination; Other: 24 hours drug withdrawal of dopaminergic medication
- AMC PARK-Parkin/PARK-PINK1: Asymptomatic mutation carriers (SMC) of the Parkin or PINK1 genes will be examined.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Other: Video-based clinical examination
- Control group: A healthy control group will be examined.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Other: Video-based clinical examination

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — TMS over the left primary motor cortex will be performed. To investigate sensorimotor integration, an electrical stimulus on the right index finger will precede the TMS pulse.
Other: Video-based clinical examination — A standardized neurological examination will be performed and video taped. The videos will be rated by movement disorder specialists, wo are blinded for the symptom and mutation status of the participants.
Other: 24 hours drug withdrawal of dopaminergic medication — Examinations will be done under chronic dopaminergic treatment and after a 24 hours dopaminergic drug withdrawal.
  Groups: SMC DYT/PARK-GCH1; SMC DYT/PARK-TAF1; SMC PARK-Parkin/PARK-PINK1
Other: Evaluation of deep brain stimulation — Examinations will be done before and after implantation of deep brain stimulation (clinically optimal stimulation vs. switched off stimulation)
  Groups: SMC DYT/PARK-TAF1

SUMMARY:
Hereditary Parkinson and dystonia syndromes are rare, as are people who carry the predisposition for Parkinson or dystonia but do not have symptoms. It is particularly important to study these people because they are a good model for understanding the development of common non-hereditary Parkinson's and dystonia. To do this, the investigators want to look at how the brain works and how different areas of the brain communicate with each other. The investigators want to identify differences in brain regions connecting perception and action between mutation carriers that develop clinical symptoms and those who stay healthy in different subgroups of inherited Parkinson-dystonia syndromes. Mutation carriers with and without symptoms of three different inherited Parkinson-dystonia syndromes will be investigated at their homes with the help of a mobile examination unit. To detect even subtle signs, which the mutation carriers might not even be aware of, the investigators will use a detailed video-based and -documented movement examination and a non-invasive magnetic stimulation technique that investigates how a sensory, i.e., electrical stimulus can influence the motor response in a hand muscle. Our study will allow the investigators, on the one hand, to define specific markers that protect some mutation carriers from having clinical symptoms and, on the other hand, to identify neurophysiological characteristics that all mutation carriers share whether or not they have clinical symptoms. These are important information for a better understanding of the basis of these disorders and for the development of new treatment strategies, which can also be transferred to genetically-undefined Parkinson's and dystonia syndromes. Through this study, large groups of mutation carriers that have received an in-depth clinical and neurophysiological examination and can be investigated longitudinally in future studies will be build up.

DETAILED DESCRIPTION:
Monogenic Parkinson-dystonia syndromes are rare but very valuable model disorders for genetically undefined syndromes, as their genetic cause, i.e., pathogenic gene variants, have been identified. For certain subtypes, even the neuroanatomical basis was discovered. Despite the different genetic and anatomical characteristics, a strong clinical overlap was reported between PARK-Parkin/PARK-PINK1, DYT/PARK-GCH1, and DYT/PARK-TAF1.

Interestingly, previous research in these different Parkinson-dystonia syndromes suggests a distinct pattern of neurophysiological alterations within the primary motor and premotor-motor network for each syndrome. Even asymptomatic, heterozygous mutation carriers, show abnormalities within neurophysiological and in addition, functional, metabolic, and structural imaging studies.

In general, a better clinical and neurophysiological evaluation of asymptomatic compared to symptomatic mutation carriers and healthy controls across subgroups is warranted. However, the number of mutation carriers per subgroup is limited and some are unable to travel to Lübeck to participate in research. To increase the participant size, in addition to the examination in our neurophysiological laboratory, the investigators want to visit and investigate some mutation carriers in their home environment with a mobile examination unit. In this regard, the transcranial magnetic stimulation paradigm of short-latency afferent inhibition (SAI) is of great interest as it can reliably capture the effects of sensory input (median nerve stimulation) on motor output (MEP amplitude) without complex neuronavigation. Additionally, a video-based clinical examination will be performed, which will be rated offline in a blinded fashion by movement disorder specialists to correlate SAI with symptom severity.

Therefore, the proposed project will, for the first time, allow a direct comparison of sensorimotor integration deficits in correlation to clinical signs between three different monogenic Parkinson-dystonia syndromes. Furthermore, contrasting the findings between asymptomatic and symptomatic mutation carriers will help, on the one hand, to draw conclusions on potential protective markers, and on the other hand, to identify neurophysiological endophenotypes. Furthermore, successful completion of the project will generate clinically well-defined monogenic subgroups with particular sensorimotor abnormalities, who can serve as model disorders in further research projects that aim to characterize sensorimotor deficit in a cognitive framework and in a longitudinal fashion.

ELIGIBILITY:
Inclusion criteria for mutation carriers:

* Pathogenic Parkin, PINK1, GCH1, or TAF1 gene variant
* Age >18 years
* Informed consent

Inclusion criteria for healthy control participants:

* No movement disorder
* Age >18 years
* Informed consent
* No medication with influences on the central nervous system

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Epilepsy
* Medication that reduces the seizure threshold

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will include symptomatic and asymptomatic carriers of pathogenic variants in the Parkin, PINK1, GCH1, or TAF1 gene, and sex- and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Contrast sensorimotor integration in patients with three different monogenic Parkinson-dystonia syndromes. | Two timepoints (if applicable): With chronic dopaminergic medication vs. 24h drug withdrawal OR before and after deep brain stimulation implantation
  Transcranial magnetic stimulation (short-latency afferent inhibition)
Define whether asymptomatic mutation carriers show abnormalities in sensorimotor integration and clinical signs of Parkinson and dystonia upon video examination. | One timepoint
  Video based clinical examination
Correlate clinical symptom severity with changes in sensorimotor integration. | Two timepoints (patients) or one timepoint (asymptomatic mutation carriers and healthy control participants)
  Transcranial magnetic stimulation (short-latency afferent inhibition) and Video based clinical examination
Evaluate treatment effects on sensorimotor integration, e.g., for PARK-Parkin/PARK-PINK1 and DYT/PARK-GCH1 chronic dopaminergic medication and for DYT/PARK-TAF1 deep brain stimulation effects. | Two timepoints (if applicable): With chronic dopaminergic medication vs. 24h drug withdrawal OR before and after deep brain stimulation implantation
  Transcranial magnetic stimulation (short-latency afferent inhibition)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Weissbach, MD, Principal Investigator — Institute of Systems Motor Science
Locations (1):
- Institute of Systems Motor Science Lübeck, Lübeck, Schleswig-Holstein, Germany